CLINICAL TRIAL: NCT07197034
Title: A Phase 3, Multicenter, Open-Label Extension Study to Assess the Safety and Efficacy of ARD-101 in Patients With Prader-Willi Syndrome
Brief Title: The Hunger Elimination or Reduction Objective (HERO ) Open -Label Extension (OLE) Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aardvark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVK-101-302
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Hyperphagia; Prader-Willi Syndrome; Hyperphagia in Prader-Willi Syndrome
Keywords: Prader-Willi Syndrome; ARD-101; PWS; Prader-Willi; Prader Willi; Prader Willi Syndrome
MeSH Terms: conditions — Hyperphagia; Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARD-101 (Experimental): (Open-label)
  Interventions: Drug: ARD-101

INTERVENTIONS:
Drug: ARD-101 — 200 mg BID (twice per day) for 1 week, 400 mg BID for 1 week, 800 mg BID for 50 weeks

SUMMARY:
The goal of this clinical trial is to learn if ARD-101 works to treat hyperphagia-related behavior in patients with Prader-Willi syndrome (PWS) when used in a long term setting. It will also teach us about the safety of ARD-101.

The main questions it aims to answer are:

What medical problems do participants have when taking ARD-101 in a long term setting

Does ARD-101 improve the total score of the HQCT-9 (hyperphagia questionnaire for clinical trials, 9 questions)?

Eligible participants will:

Have completed treatment on the AVK-101-301 study through Week 12/End of Treatment

Take ARD-101 every day for up to 12 months.

Visit the clinic at Months 1, 3, 6 and 12 during dosing and then have tele-visits at Week 2, Months 3 and 9, then 4 weeks after stopping the ARD-101.

Patients/Caregivers will keep a daily diary.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed treatment on Aardvark Therapeutics clinical study AVK-101-301

Exclusion Criteria:

* Any complications that makes participation unsafe in the Investigator's opinion

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in Hyperphagia Questionnaire for Clinical Trials (HQ-CT) Score | During treatment period (approximately 12 months)
  The HQ-CT score is a 9 question, 5-point scale to describe the PWS patient's hyperphagia food-related problem behaviors. It is completed by the patient's caregiver. Each question is scored from 0 to 4. The minimum total score is 0 (hyperphagia related behavior symptoms not exhibited) and the maximum total score is 36 (hyperphagia related behavior symptoms are observed).

SECONDARY OUTCOMES:
Change in Caregiver Global Impression of Severity (CaGI-S) for Hyperphagia in Prader-Willi patients | During treatment period (approximately 12 months)
  The CaGI-S is a single-item, 7-point scale to describe the severity of the PWS patient's hyperphagia (excessive hunger). It is completed by the patient's caregiver. The minimum score is 1 (not present) and the maximum score is 7 (extremely severe). A higher score indicates a worse severity of hyperphagia.

CONTACTS AND LOCATIONS:
Locations (42):
- United States (15):
  - Children's of Alabama, Birmingham, Alabama
  - Stanford Children's Health Specialty Services, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado, Denver, Colorado
  - Nemours Children's Clinic Wilmington, Wilmington, Delaware
  - UF Shands Children's Hospital, Gainesville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Children's Ambulatory Care Center, Mineola, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
- Canada (3):
  - Alberta Children's Hospital Research Institute, Calgary, Alberta
  - Li Ka Shing Centre for Health Research Innovation, Edmonton, Alberta
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- France (5):
  - CHU de Toulouse-Hôpital Des Enfants, Toulouse, Haute-Garonne
  - CHU d'Angers, Angers, Maine-et-Loire
  - AP-HP - Hôpital de la Pitié Salpétrière, Paris
  - AP-HP - Hôpital universitaire Necker-Enfants malades, Paris
  - CHU de Toulouse- Hôpital de Rangueil, Toulouse
- Italy (3):
  - Ospedale Pediatrico Bambino Gesù IRCCS, Rome, Lazio
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Florence, Tuscany
- Romania (3):
  - National University Hospital for Children's Neurorehabilitation "Dr. Nicolae Robanescu", Bucharest, București
  - Institutul National de Endocrinologie C. I. Parhon, Bucharest
  - Spitalul Clinic de Urgenta Sfantul Spiridon, Iași
- South Korea (3):
  - Inha University Hospital, Incheon
  - Samsung Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (3):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (4):
  - Fulborn Hospital, Cambridge
  - Royal Hospital for Children (Glasgow) - PPDS - PIN, Glasgow
  - Leicester Royal Infirmary, Leicester
  - The Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: No